CLINICAL TRIAL: NCT02842047
Title: Self-Management of Stress in Caregivers of Cancer Patients
Brief Title: The Mediating Effects of Decentering on Self-Management of Stress and End of Life Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4815
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Stage IV Gastrointestinal Cancer; Advanced Gynecological Cancer
Keywords: caregiver; end of life
MeSH Terms: conditions — Gastrointestinal Neoplasms; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End of Life Care with Meditation (Experimental): The intervention has two content components: end of life planning education (using end of life planning videos) and strategies and kindness based meditation (using the Stop, Breathe & Think™ app). The activities comprising these components work together to improve both analytic neural processing (e.g. improving knowledge about goal setting and EOL planning, learning self-monitoring of EOL values and goals of care, and self-regulation skills of monitoring symptoms of distress and anxiety) and emotional neural processing (e.g. teaching participants to experience the moment non-judgmentally and directing thoughts to think positive thoughts and feel positive feelings like kindness and compassion.
  Interventions: Behavioral: Stop, Breathe & Think™; Behavioral: End of Life Planning Videos
- Meditation Only (Active Comparator): This arm has the single content component of kindness based meditation delivered by using the Stop, Breathe & Think™ application. This group will also be instructed to view 3 caregiver wellness videos.
  Interventions: Behavioral: Stop, Breathe & Think™; Behavioral: Caregiver wellness videos

INTERVENTIONS:
Behavioral: Stop, Breathe & Think™ — online daily meditations delivered using smart phone or other computer based application
  Other Names: meditation app
Behavioral: End of Life Planning Videos — Three videos, each 10 minutes in length which will be viewed over the study period. The videos will walk participants though key aspects of end of life planning.
  Other Names: online videos
  Arms: End of Life Care with Meditation
Behavioral: Caregiver wellness videos — Three videos, each 10 minutes in length which will be viewed over the study period. The videos will walk participants though general caregiver wellness.
  Arms: Meditation Only

SUMMARY:
Caregivers of persons with cancer may face many challenges as they support and care for a person receiving treatment. Sometimes having to help make treatment decisions for a patient can cause distress for caregivers. The purpose of this study is to evaluate 2 different electronic approaches to providing support for a caregiver. One group will have access to an on-line program with videos, providing education on decision making strategies for caregivers of patients with cancer, to watch and a daily meditation application and the other group will have access to the daily meditation application. Investigators will randomly assign participants to each group.

DETAILED DESCRIPTION:
Investigators will conduct a randomized trial pilot study to examine two arms of the intervention among 20 caregivers of patients with advanced cancer. Investigators will collect mixed methods data to describe changes in proximal and distal outcomes. Investigators have chosen the time points to capture neural and behavioral changes associated with the intervention and to capture end of life quality of life (QOL) for a majority of caregivers after death of their loved one. Investigators aim to:

1. Evaluate the short and longer-term effects of the end of life care with medication (EOL_M) and meditation only (M_Only) interventions on stress reduction and end of life (EOL) planning behaviors and determine if there are different effects between EOL_M and M_ Only interventions.
2. Evaluate the short-term and long-term effects of the intervention on caregiver distress, decisional regret, and EOL values and goals of care for treatment.
3. Evaluate the impact of decentering on the association between the interventions, self-management behaviors (stress reduction and EOL planning behaviors) and distress, anxiety, concordance between EOL values and goals of care for treatment, decisional regret and satisfaction with EOL care.
4. Describe the neural activity processes that are associated with increased self-management activities.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of patients who have been diagnosed with Stage IV gastrointestinal (GI) cancer
* coming with the patient at the Seidman Comprehensive Cancer Center at University Hospitals Case Medical Center (UHCMC)
* have access to the internet and a computer, tablet, or smart phone, and
* speak and comprehend English.

Exclusion Criteria:

* currently practicing mindfulness-based interventions (yoga, meditation, deep breathing)
* require psychotherapy within the last three months
* have a history of dementia, major neurological illness
* pregnant
* history of a medical condition or procedure that is contraindicated for functional magnetic resonance imaging (fMRI) scanning (i.e. cardiac pacemaker, sternal wires, or metal implants); and
* claustrophobia requiring anxiolytics or sedation; or
* expect to relocate from Northeast, Ohio within 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Repeated Measures ANCOVA Model (F-Statistic) | At 10 months
  Estimation of effect of the intervention
Repeated Measures ANCOVA Model (F-Statistic) | At 1 month
  Estimation of effect of the intervention

SECONDARY OUTCOMES:
Change in National Comprehensive Cancer Network (NCNN) Distress Thermometer Score | From baseline to up to 10 months
  Measure of caregiver distress
Change in Degner's Decisional Control Scale | From baseline to up to 10 months
  Measure of decisional control
Change in End of Life Value | From baseline to up to 10 months
  Measure of end of life values and focus of care
Change in PROMIS-29 Scale | From baseline to up to 10 months
  Measure of caregiver anxiety
Change in O'Connor's Decisional Regret Scale | From baseline to up to 10 months
  Measure of decisional regret
Change in FAMCARE Scale | From baseline to up to 10 months
  Measure of satisfaction with end of life care

CONTACTS AND LOCATIONS:
Overall Officials: Sara Douglas, PhD, RN, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Moore SM, Musil CM, Alder ML, Pignatiello G, Higgins P, Webel A, Wright KD. Building a Research Data Repository for Chronic Condition Self-Management Using Harmonized Data. Nurs Res. 2020 Jul/Aug;69(4):254-263. doi: 10.1097/NNR.0000000000000435. PMID 32205788